CLINICAL TRIAL: NCT04266847
Title: Prospective Clinical Study of Preoperative and Postoperative Unilateral Mild Cataract Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20191127
Record Dates: First submitted 2019-11-29; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Cataract Senile
Keywords: unilateral cataract; binocular functional vision; Multifocal Intraocular Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- unilateral mild cataract patients (Experimental): The patients who underwent monocular IOL implantation before and then present mild cataract in the fellow eye.
  Interventions: Device: monofocal IOL,bifocal IOL,or trifocal IOL

INTERVENTIONS:
Device: monofocal IOL,bifocal IOL,or trifocal IOL — phacoemulsification and implantation of IOL.IOL may be monofocal IOL,bifocal IOL,or trifocal IOL

SUMMARY:
This is to compare preoperative and postoperative binocular functional vision in patients with unilateral intraocular len（IOL） in one eye and mild cataract in the fellow eye.

DETAILED DESCRIPTION:
The subjects are the patients who underwent monocular IOL implantation before and present mild cataract in the fellow eye.Compare preoperative and postoperative the binocular functional vision and the satisfaction of patients when the patients ask for the surgery (phacoemulsification and IOLs implantation)on the fellow eye. The type of IOLs maybe according to the patients preference and the eyes condition.The subjects will be divided into three groups according to the type of the IOLs，including monofocal group,bifocal group,and trifocal group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had monocular intraocular lens in one eye with mild cataract in the fellow eye ask for the cataract surgery in the fellow eye
* Regular corneal topography and corneal astigmatism ≤ 0.75 Diopter

Exclusion Criteria:

* Pregnant or nursing women
* In the presence of other ocular diseases that may affect the stability of the lens capsule (pseudoexfoliation syndrome, glaucoma, traumatic cataract, Marfan syndrome, etc.)
* In the presence of other ocular diseases that is expected to have a poor final visual acuity of worse than 0.2 logMAR after surgery (amblyopia, strabismus, keratoconus, etc.)
* Pupil abnormality (non-reactive pupil, tonic pupils, abnormally shaped pupils, etc.)
* Patients using systemic or ocular medication that affect visual acuity.
* Patients with history of ocular trauma or prior ocular surgery including refractive procedures
* Patients participating in other clinical trials during the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
binocular visual acuity | 3 months postoperatively
  uncorrected distance visual acuity (UCVA), intermediate visual acuity, near visual acuity will be measured at 5m, 80cm and 40cm respectively. All visual acuity measurements will be conducted under photopic conditions (85 cd/m2) and at 100% contrast

SECONDARY OUTCOMES:
Binocular Contrast sensitivity | 3 months postoperatively
  Contrast sensitivity measures will be conducted binocularly, under photopic, mesopic (5 cd/m2), photopic with glare and mesopic with glare conditions, with the OPTEC 6500 contrast sensitivity test (Stereo Optical, USA). Contrast sensitivity will be evaluated at five spatial frequencies (1.5, 3, 6, 12, and 18 cycles per degree [cpd]). Patients will be allowed 5 minutes to adapt to each illumination level before testing
Binocular Defocus Curve | 3 months postoperatively
  Binocular defocus curves will be obtained in all patients, positioned at 5m under photopic (>85 cd/m 2 ) condition to measure the visual acuity with each defocus lens, representing the consecutive visual function of each eye. Negative lenses were added in 0.50 D steps and the visual acuity will be recorded for each type of defocus level. The procedure will be then repeated but with positive lenses. The range of defocus evaluated is from -4.00D to +2.00D.
stereopsis | 3 months postoperatively
  Use block diagram of random-spot synoptophore to observe long distance stereopsis vision and yan's stereogram to observe short distance stereopsis vision.
Fusion function | 3 months postoperatively
  The fusion function of perception and movement (convergence and divergence)will be examined with a synoptophore.
Subjective visual quality | 3 months postoperatively
  Photic phenomena (score according to severity,0~4, higher scores mean worse)and spectacle dependence percentages will be evaluated by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Hong, PhD，MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No